CLINICAL TRIAL: NCT04787835
Title: The Effect of Forearm Nerve Blocks on Pain-free Tourniquet Time Compared to Local Anesthetic for Awake Hand Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Christian Petropolis, Assistant professor and Residency Program Director, Department of Surgery, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2021:003
Record Dates: First submitted 2021-03-02; First posted 2021-03-09 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Fracture Fixation, Internal; Metacarpal Fracture; Finger Fracture; Anesthesia, Local; Tendon Injury - Hand
Keywords: Anesthesia, local; Minor surgical procedure; Hand injuries
MeSH Terms: conditions — Hand Injuries

STUDY DESIGN:
Intervention Model Description: Patients who consent to participation will then be randomized using a random number generator to receive either a forearm nerve block or local anesthetic infiltration, there will be 20 patients assigned to each group.
Masking Description: The study will be open-label as both the patient and resident/surgeon will be aware of the type of block (forearm vs local) performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Forearm Nerve Block (Experimental): Patients will receive a nerve block of the radial, median, and ulnar nerves at the level of the forearm using 1% lidocaine with epinephrine. The lidocaine will be injected subcutaneously, using a total dose of less than 7mg per kilogram.
  Interventions: Procedure: Forearm nerve block
- Local Anesthetic Infiltration (Active Comparator): Patients will receive local anesthetic infiltration, using 1% lidocaine with epinephrine, to the fracture site and surrounding tissue. No nerve blocks will be performed. The lidocaine will be injected subcutaneously, using a total dose of less than 7mg per kilogram.
  Interventions: Procedure: Local anesthetic infiltration

INTERVENTIONS:
Procedure: Forearm nerve block — Local anesthesia will be used to perform a forearm block of the median, radial, and ulnar nerves.
  Arms: Forearm Nerve Block
Procedure: Local anesthetic infiltration — Local anesthesia will be infiltrated at the site of injury
  Arms: Local Anesthetic Infiltration

SUMMARY:
Wide-awake surgery with local anesthesia is a widely described approach to performing numerous minor hand procedures, such as tendon repairs and percutaneous fracture pinning, but is less frequently used for longer procedures such as open reduction internal fixation (ORIF). This is in part due to the need for a tourniquet for improved visualization, however pain-free tourniquet time with local anesthesia is roughly 20 minutes, shorter than the average time for ORIFs (Gillis), for example. While general anesthesia may still be avoided with more proximal blocks such as a brachial plexus or bier blocks, these still require presence of an anesthesiologist during the procedure, increasing human resource utilization and costs. Development of an anesthetic technique for hand surgery which could be performed by surgeons in a clinic setting, that still provides sufficiently long pain-free tourniquet times could decreases costs and wait times.

The investigators hypothesize that the pain patients experience after 20 minutes of tourniquet application with local anesthetic infiltration is not due to direct pressure on the proximal arm, but rather distal digital ischemia pain. Previously, it has been shown that ultrasound-guided regional block of the median, radial, and ulnar nerves in the forearm is effective analgesia for awake hand surgery (Winter).

Currently, there are no randomized studies investigating if forearm nerve blocks can prolong pain-free tourniquet time compared to local anesthesia infiltration, by blocking this ischemic pain in the distal arm. The investigators' objective is therefore to determine if forearm nerve blocks prolong pain-free tourniquet time compared to local anesthetic infiltration.

DETAILED DESCRIPTION:
With increasing caseloads in some healthcare systems, patients requiring hand surgery may wait over two weeks for time in the general operating room schedule. During this time, fractures may heal, or tendons may retract, leading to a need for more extensive and longer procedures such as osteotomies or tendon reconstruction. It also prolongs time away from work, as well as home for rural patients who must relocate while awaiting surgery in major centers. Previously, it has been shown that performing closed hand fracture fixation on awake patients in a clinic or procedure room setting leads to 60-100% increases in daily case volume compared to the main operating room (OR) (Gillis, Steve). Fixation of hand fractures in this setting has also been shown to cost over 2000$ less than in the OR, by reducing staffing requirements, equipment, and anesthesia costs (Steve).

Performing hand surgery in awake patients under local anesthesia has been shown by numerous studies to be a safe and effective. Wide-awake hand surgery is generally well-tolerated, has lower post-operative opioid requirements, and is often preferred by patients (Thompson). Furthermore, by preventing the need for general anesthesia, this technique allows hand surgery to be performed in patients who may otherwise not be operative candidates. During flexor tendon repair, awake surgery provides the unique advantage of being able to actively test the repair intraoperatively. In Canada, awake surgery under local anesthesia is commonly done for tendon repairs, carpal tunnel release, and percutaneous pinning of fractures without a tourniquet (Gillis, Steve, Peters). While tourniquet use improves visualization of the operative field, when only local anesthesia is used patients can typically tolerate the tourniquet for less than 20 minutes before pain begins.

However, for ORIFs, flexor tendon repairs, etc., the use of a tourniquet is ideal for exposure of the operative site. Current literature suggests that the maximum pain-free tourniquet time is roughly 20 minutes, which is less than the average length of ORIFs (Gillis) and flexor tendon repair. Intravenous regional anesthesia (IVRA), i.e. Bier blocks, are well-established means of providing anesthesia for hand surgeries requiring tourniquet use, and enable tourniquet times from 20 minutes to two hours (Dekoninck, Brown). While these blocks prevent the need for general anesthesia, they still require an anesthetist to perform and monitor the block. More recently, forearm tourniquets with IVRA have been shown to be non-inferior to traditional proximal arm tourniquets, with lower doses of post-operative opioids required (Dekoninck, Farbood). However, compared to local anesthesia, IVRA for procedures were tourniquets are preferred still increases costs, staffing requirements, and resource use as they often take place in the OR. However, local anesthetic infiltration by the treating surgeon may not provide sufficient pain relief for the amount of tourniquet time required to complete many hand surgeries. Therefore, although many methods of anesthesia for hand surgery exist, include local anesthetic infiltration and proximal nerve blocks, there is not yet one 'gold standard' approach.

Ultrasound guided peripheral nerve blocks at the forearm level have previously been shown to be a safe, effective method of providing regional anesthesia for minor hand procedures, that are tolerated well by patients (Winter). The technique can be quickly taught to even junior residents, and does not require any specialized equipment outside of the ultrasound probe (Winter). These blocks take roughly five minutes to perform, and anesthesia is achieved after an additional five minutes, shorter than typical times for blind forearm nerve blocks (Lovely).

The investigators hypothesize that the pain patients experience after 20 minutes of tourniquet application with local anesthetic infiltration is not due to direct pressure on the proximal arm, but rather distal digital ischemia pain. Previously, it has been shown that ultrasound-guided regional block of the median, radial, and ulnar nerves in the forearm is effective analgesia for awake hand surgery (Winter). Currently, there are no randomized studies investigating if forearm nerve blocks can prolong pain-free tourniquet time compared to local anesthesia infiltration, by blocking this ischemic pain in the distal arm. The investigator's aim is therefore to determine if forearm nerve blocks prolong pain-free tourniquet time compared to local anesthetic infiltration.

All patients over 18 years of age, booked for an awake hand surgery will be considered for inclusion. These patients will be identified through emergency room consults, referrals from outside centers, and attending surgeon clinics at our institution. Currently, if patients require minor hand surgeries, they are then assessed for suitability for having their procedure while awake using local anesthesia. Patients who are candidates for awake surgery will then be informed of the research study by a resident, physician assistant, or attending physician, and have the opportunity to consent to participation. This will not be done by a resident/physician assistant/attending physician who will be performing or assisting with the procedure. Patients who consent to participation will then be randomized using a random number generator to receive either a forearm nerve block or local anesthetic infiltration. The study will be open-label as both the patient and resident/surgeon will be aware of the type of block (forearm vs local) performed.

The risks and benefits associated with forearm and local anesthesia blocks will be explained to the patient as part of the informed consent, prior to randomization. Patients will be recruited from attending physician clinics, however the staff screening patients for eligibility and conducting informed consent will not be the individual who is either a) performing the surgery, or b) collecting, analyzing, or interpreting the data. Patients will have the remaining length of their clinic appointment to contemplate participation in the study.

If patients in either group begin to experience pain during their procedure the tourniquet will be taken down and the time will be recorded. Participants in both groups will receive adequate analgesia, as additional local anesthetic will be administered if patients express pain during the procedure. Total procedure time will also be recorded.

The resident/physician performing the procedure will record the patient's diagnosis, type of procedure, location, duration of the entire procedure, type and amount of local anesthetic used, and duration of pain-free tourniquet time. Any additional local anesthetic required during the procedure will be recorded. Any deviations from the expected procedure, or intraoperative complications will also be recorded. The REB will be notified of any harms to patients, as a result of the study, occur. Any subsequent recommendations from the REB regarding study termination will be followed. If any patients experience local anesthetic toxicity, sustain nerve or blood vessel damage, or experience other intraoperative complications as a result the study intervention(s), the study will be placed on hold until full review of the data is complete, and terminated if appropriate. Patients who were involved of the study to date will be contacted explaining the reason for termination of the study.

After the procedure, the resident involved in the procedure will provide the patient with the survey questions. The individuals conducting the surveys will not otherwise be involved in the study. This will be a two question survey recording the amount of pain felt during the procedure and overall experience with their awake hand surgery. Both questions will be scored on a Numerical analogue scale (NAS) from 1-10. If the patient is unable to physical write due to splinting of the dominant hand, the resident will record the answers verbalized by the patient.

Data from the study will be reviewed on a weekly basis. All complications will be noted. Any major complication (resulting in harm or near-harm to a patient) will prompt review of the study data to date for any further complications, including which group the participant(s) experiencing the complication were assigned to.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* 18 years of age or older at time of enrollment
* are scheduled to undergo a minor hand surgery under local anesthesia

Exclusion Criteria:

* Patients with known allergies or intolerance to local anesthetic agents
* Patients with known chronic pain disorders or peripheral neuropathies
* Pediatric patients (<18 years of age) at the time of enrollment
* Patients with a history of opioid (or other pain medication) substance use disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Pain-free tourniquet time (minutes) | Pain-free tourniquet time; from the time of tourniquet inflation until the patient experiences tourniquet pain, whichever occurs first
  When upper extremity surgery is performed with local anesthesia and a tourniquet, the tourniquet must be removed after roughly 20 minutes as patients begin to feel tingling and pain in their hand.
  Pain-free tourniquet time refers to the amount of time the tourniquet is applied before the patient begins to feel an uncomfortable sensation or pain in the arm to which the tourniquet is applied. Once pain occurs the tourniquet is released. This will be measured in minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Petropolis, MD, Principal Investigator — University of Manitoba

IPD SHARING:
Plan to Share IPD: Yes
We do intend to make individual participant data (IPD) data available to other researchers upon completion of the study. This includes information related to the primary outcome (pain-free tourniquet time) as well as participant responses to our post-procedure questionnaire, which contains a subjective rating of pain and overall experience during the procedure on a numeric scale.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Information will be made available from the end of the study period, for one calendar year after publication of our results, upon request.
Access Criteria: We are currently working with our institutional library to formalize how this data will be shared.

REFERENCES:
- [Background] Feehan LM, Sheps SB. Incidence and demographics of hand fractures in British Columbia, Canada: a population-based study. J Hand Surg Am. 2006 Sep;31(7):1068-74. doi: 10.1016/j.jhsa.2006.06.006. PMID 16945705
- [Background] Gillis JA, Williams JG. Cost analysis of percutaneous fixation of hand fractures in the main operating room versus the ambulatory setting. J Plast Reconstr Aesthet Surg. 2017 Aug;70(8):1044-1050. doi: 10.1016/j.bjps.2017.05.011. Epub 2017 May 20. PMID 28572044
- [Background] Steve AK, Schrag CH, Kuo A, Harrop AR. Metacarpal Fracture Fixation in a Minor Surgery Setting Versus Main Operating Room: A Cost-minimization Analysis. Plast Reconstr Surg Glob Open. 2019 Jul 5;7(7):e2298. doi: 10.1097/GOX.0000000000002298. eCollection 2019 Jul. PMID 31942336
- [Background] Thompson NB, Calandruccio JH. Hand Surgery in the Ambulatory Surgery Center. Orthop Clin North Am. 2018 Jan;49(1):69-72. doi: 10.1016/j.ocl.2017.08.009. PMID 29145986
- [Background] Peters B, Giuffre JL. Canadian Trends in Carpal Tunnel Surgery. J Hand Surg Am. 2018 Nov;43(11):1035.e1-1035.e8. doi: 10.1016/j.jhsa.2018.02.014. Epub 2018 Mar 17. PMID 29559326
- [Background] Dekoninck V, Hoydonckx Y, Van de Velde M, Ory JP, Dubois J, Jamaer L, Jalil H, Stessel B. The analgesic efficacy of intravenous regional anesthesia with a forearm versus conventional upper arm tourniquet: a systematic review. BMC Anesthesiol. 2018 Jul 18;18(1):86. doi: 10.1186/s12871-018-0550-4. PMID 30021514
- [Background] Brown EM, McGriff JT, Malinowski RW. Intravenous regional anaesthesia (Bier block): review of 20 years' experience. Can J Anaesth. 1989 May;36(3 Pt 1):307-10. doi: 10.1007/BF03010770. PMID 2720868
- [Background] Farbood A, Khademi S, Tajvidi R, Hooshangi M, Salari S, Ghani M, Tahmasebi S, Jamali H. Comparison of Intravenous Regional Anesthesia with Single-Cuff Forearm Tourniquet and Hematoma Block and Traditional Method in Patients with Distal Radius Fractures; A Randomized Clinical Trial. Bull Emerg Trauma. 2020 Apr;8(2):77-82. doi: 10.30476/BEAT.2020.46446. PMID 32420391
- [Background] Winter J, McLeod G, Quaife T, Petropolis C. Surgeon-administered Ultrasound-guided Peripheral Nerve Blocks in Outpatient Procedures of the Upper Extremity. Plast Reconstr Surg Glob Open. 2020 Nov 24;8(11):e3227. doi: 10.1097/GOX.0000000000003227. eCollection 2020 Nov. PMID 33299698
- [Background] Lovely LM, Chishti YZ, Woodland JL, Lalonde DH. How Much Volume of Local Anesthesia and How Long Should You Wait After Injection for an Effective Wrist Median Nerve Block? Hand (N Y). 2018 May;13(3):281-284. doi: 10.1177/1558944717709072. Epub 2017 May 26. PMID 28549398